CLINICAL TRIAL: NCT02944955
Title: A Study of BLEX 404 Oral Liquid in Patients With International Prognostic Scoring System (IPSS) Intermediate-1, Intermediate-2 or High-Risk Myelodysplastic Syndrome (MDS) and Chronic Myelomonocytic Leukemia (CMML)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI-1301-01
Record Dates: First submitted 2016-10-04; First posted 2016-10-26 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BLEX 404 Oral Liquid (Experimental): Part I:
  Part I-1: Low Dose BLEX 404 Oral Liquid (3 mg/kg, BID) is administered in combination with 2 cycles of azacitidine.
  Part I-2: High Dose BLEX 404 Oral Liquid (4.5 mg/kg, BID) is administered in combination with 2 cycles of azacitidine.
  Part II:
  Recommended Dose Level (RDL) of BLEX 404 Oral Liquid will be determined by results from Part I.
  BLEX 404 Oral Liquid at RDL is administered in combination with 6 cycles of azacitidine.
  Interventions: Drug: BLEX 404 Oral Liquid

INTERVENTIONS:
Drug: BLEX 404 Oral Liquid — BLEX 404 Oral Liquid is orally administered twice daily in combination with azacitdine treatment cycles (2 cycles in Part I and 6 cycles in Part II).
  Azacitidine treatment: SC or IV injections at 75 mg/m2, QD for 7 days each cycle. 28 days/cycle, and repeat cycles every 4 weeks.

SUMMARY:
This is a clinical trial to determine the safety, recommended dose level (RDL), and infection control of BLEX 404 Oral Liquid in combination with azacitidine in patients with International Prognostic Scoring System (IPSS) intermediate-1 (int-1), intermediate-2 (int-2) or high-risk myelodysplastic syndrome (MDS) and Chronic Myelomonocytic Leukemia (CMML).

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or older, able to sign informed consent, understand and comply with protocol requirements and instructions.
* Body weight between 30 to 120 kg
* International Prognostic Scoring System (IPSS) intermediate-1 (int-1), intermediate-2 (int-2) or high-risk myelodysplastic syndrome (MDS) by World Health Organization (WHO) or Chronic Myelomonocytic Leukemia (CMML) patients.
* Not previously treated with MDS and CMML therapy and require treatment with azacitidine* for the first time at 75 mg/m2 subcutaneously or intravenously, daily for 7 days (7 nonconsecutive day of 6-1-1 or 5-2-2 treatment schedule is acceptable in which the drug is administered Monday-Saturday and then Monday of the following week for a 6-1-1 schedule, and in which the drug is administered Monday-Friday and then Monday-Tuesday of the following week for 5-2-2 schedule) per cycle. Treatment of the study drug, BLEX 404 Oral Liquid will begin at the same time receiving the first dose of azacitidine in this study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-3.
* Adequate baseline organ function defined by the criteria below: total bilirubin ≤ 1.5x the upper limit of normal (ULN) except for Gilbert's syndrome or indirect hyperbilirubinemia due to hemolysis; ALT ≤ 2.5x ULN; AST ≤ 2.5x ULN; creatinine clearance ≥ 60 mL/min/1.73 m2.
* Women must be either of non-child bearing potential, or women with child-bearing potential and men with reproductive potential and a female partner of childbearing potential must either have had a prior vasectomy or agree to use effective contraception from time of Screening Visit until the Follow-Up Visit.

Exclusion Criteria:

* Historical allergic events caused by mushroom.
* Previous treatment with hypomethylating agent or known immediate or delayed hypersensitivity reaction to drugs chemically related to azacitidine that contraindicates the subjects' participation.
* Patients with active infections or require treatments with immunosuppressive drugs at screening visit. However, patients require ongoing treatments with corticosteroids may be recruited.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of BLEX 404 Oral Liquid.
* Any serious and/or unstable pre-existing medical condition (including any advanced malignancy other than the disease under study), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures.
* Any clinically significant pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal or genitourinary disease unrelated to underlying hematologic disorder.
* Active and uncontrolled infections of the following: hepatitis B (HBV), hepatitis C (HCV), and human immunodeficiency virus (HIV) infection. However, HBV and HCV carriers with viral load test of "not detected" or "negative" results may be recruited in this study.
* Lactating female and women with a positive serum or urine pregnancy test at screening assessments.
* (For Part II Interventional Study subjects only) No indication, in the opinion of the treating physician, for antibiotic prophylaxis within 2 weeks prior to study treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Part I: Recommended dose level (RDL) of BLEX 404 Oral Liquid | 8 weeks (2 cycles of azacitidine)
  RDL is defined by BLEX 404 Oral Liquid-related prohibited toxicity in subjects undergoing 2 cycles of azacitidine treatment. When one of the stopping criteria is met during the study treatment period, RDL will be set at the lower dose level.
Part II: Incidence of infections | 24 weeks (6 cycles of azacitidine)
  Number of subjects experience infection events and inpatient hospitalization due to infections.

SECONDARY OUTCOMES:
Part I: (A) Number of subjects experience infections events and inpatient hospitalization due to infections | 8 weeks (2 cycles of azacitidine)
Part I: (B) Treatments and duration of each infections | 8 weeks (2 cycles of azacitidine)
Part I: (C) Complete remission (CR) or partial remission (PR) of bone marrow, peripheral blood, cytogenetic response (defined by 2006 IWG Criteria) | 8 weeks (2 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 2 cycles of azacitidine.
Part I: (D) Hematological improvement of erythroid (hemoglobin and RBC-transfusion independence), neutrophil (Absolute Neutrophil Count), and platelet (platelet count) response (defined by 2006 IWG Criteria) | 8 weeks (2 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 2 cycles of azacitidine.
Part I: (E) Frequency and requirement of red blood cell transfusion (defined by 2006 IWG Criteria) | 8 weeks (2 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 2 cycles of azacitidine.
Part I: (F) Disease Progression (defined by 2006 IWG Criteria) | 8 weeks (2 cycles of azacitidine)
  Disease progression of bone marrow, erythroid (hemoglobin and RBC-transfusion independence), and platelet (platelet count) in subjects undergone BLEX 404 Oral Liquid treatment in combination with 2 cycles of azacitidine.
Part II: (A) Time-to-first infection | 24 weeks (6 cycles of azacitidine)
Part II: (B) Duration (days) of each infection event | 24 weeks (6 cycles of azacitidine)
Part II: (C) Number of infections requiring supportive care or antimicrobial agents | 24 weeks (6 cycles of azacitidine)
Part II: (D) Duration (days) of treatments for infections | 24 weeks (6 cycles of azacitidine)
Part II: (E) Complete remission (CR) or partial remission (PR) of bone marrow, peripheral blood, cytogenetic response (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 6 cycles of azacitidine.
Part II: (F) Hematological improvement of erythroid (hemoglobin and RBC-transfusion independence), neutrophil (Absolute Neutrophil Count), and platelet (platelet count) response (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 6 cycles of azacitidine.
Part II: (G) Frequency and requirement of red blood cell transfusion (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  Hematological Response in subjects undergone BLEX 404 Oral Liquid in combination with 6 cycles of azacitidine.
Part II: (H) Disease Progression (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  Disease progression of bone marrow, erythroid (hemoglobin and RBC-transfusion independence), and platelet (platelet count) in subjects undergone BLEX 404 Oral Liquid treatment in combination with 2 cycles of azacitidine.
Part II: (I) Six-month overall survival rate (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  defined as time from beginning of treatment till death from any cause occurs or last follow-up.
Part II: (J) Six-month progression-free survival (defined by 2006 IWG Criteria) | 24 weeks (6 cycles of azacitidine)
  defined as time from beginning of treatment till disease progression, death from MDS or CMML, or last follow-up.
Part II: (K) Immune Response | 24 weeks (6 cycles of azacitidine)
  Neutrophil and monocyte function by respiratory burst assay